CLINICAL TRIAL: NCT05374200
Title: A Randomized Control Trial Evaluating the Impact of a 12-week Mind-body Wellness Intervention in Patients With Primary Biliary Cholangitis (PBC)
Brief Title: Mind-body Wellness Intervention in Primary Biliary Cholangitis (PBC)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pro00112622
Record Dates: First submitted 2022-04-01; First posted 2022-05-16 (Actual); Last update posted 2022-08-03 (Actual); Status verified 2022-07

CONDITIONS: Primary Biliary Cirrhosis
Keywords: Mind Body Therapy; Yoga; Meditation; Behavior Change; Fatigue; Quality of Life; Stress; Depression; Anxiety
MeSH Terms: conditions — Liver Cirrhosis, Biliary; Fatigue; Depression; Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant
Masking Description: Sealed envelopes
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Participants will receive the standard of care for PBC and access to the online intervention. During the intervention period, participants will also receive weekly brief (~10-minute) motivational interview style telephone check-ins.
  Interventions: Other: Mind-body intervention with 1-1 support from study personnel
- Wait list control group (No Intervention): During the 12-week wait list period, participants will receive the standard of care for PBC in addition to weekly emails with motivational messages.

INTERVENTIONS:
Other: Mind-body intervention with 1-1 support from study personnel — The multicomponent intervention will consist of the following core components: (1) A choice between three different types of low-intensity, mindful movement videos - chair fitness, standing fitness, or standing tai chi (15-30 minutes/session); (2) Breathwork and theme-of-the-week based mindfulness meditations (5-10 minutes/session); (3) A once weekly positive psychology/behavior change activity presented as a point-and-click interactive storybook within the online site; (4) A once weekly disease management tip from a PBC physician.
  Weekly brief (~10-minute) motivational interview style telephone check-ins taking place during the intervention period will be conducted by a member of the study team. During these check-ins, progress will be reviewed, motivation provided, and questions answered.
  Other Names: Mind-body intervention
  Arms: Intervention group

SUMMARY:
The investigators have designed a guided, online, multicomponent, mind-body intervention for participants with primary biliary cholangitis. The ability of the online intervention to impact the primary and secondary outcome measures will be assessed as compared to control.

DETAILED DESCRIPTION:
Persons with primary biliary cholangitis (PBC) experience significantly higher rates of fatigue, stress, anxiety, depression, and impaired health related quality of life (HRQOL) as compared to the general population. Online wellness programming ranging from physical activity to mindfulness interventions has been shown to be effective in decreasing fatigue and improving mental wellness in a variety of chronic disease populations. To date, no large-scale studies have been conducted to discern whether programming of this nature impacts measures of wellbeing in PBC.

Building upon a 12-week, online, mind-body wellness program that our team previously co-developed with the Canadian PBC Society and launched as a feasibility and acceptability trial to a group of 30 individuals with PBC, the primary aim of this research project is to carry out a randomized controlled trial to assess the efficacy of the online intervention provided with brief study follow-up phone calls performed weekly by study personnel as compared to a control arm. The ability of the online program to impact the primary outcome measure of anxiety and depression as measured by the hospital anxiety and depression scale (HADS), and a range of secondary outcomes including perceived stress, fatigue, resilience, health related quality of life, physical functioning will be assessed as compared to control.

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥ 18 years)
* Identified diagnosis of PBC
* Ability to communicate (read, write, speak) in English
* Access to an internet connected device at home.

Exclusion Criteria:

* Inability to provide informed consent
* Unsafe to participate in a low-intensity online activity program (e.g. uncontrolled angina or arrhythmia, myocardial infarction or stroke within the last 3 month, other major medical comorbidity of concern)
* Severe psychiatric disorders (HADS score >10)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2021-10-03 (Actual); Primary Completion 2022-04-09 (Actual); Study Completion 2022-04-09 (Actual)

PRIMARY OUTCOMES:
HADS Anxiety and Depression Scale | Baseline to 12 weeks
  Depression and anxiety will be measured on the Hospital Anxiety and Depression Scale. The minimum score is 0, the maximum score is 21, and higher scores indicate a worse outcome.

SECONDARY OUTCOMES:
PBC-40 | Baseline to 12 weeks
  Six PBC specific quality of life domains will be measured on the PBC-40. For each question, the minimum value is 1, the maximum value is 5, and higher scores indicates a worse outcome. The overall scoring range varies among domains.
Perceived Stress Scale | 12 Weeks
  The degree to which situations in one's life are appraised as stressful will be assessed using the Perceived Stress Scale. The minimum score is 0, the maximum score is 40, and higher scores indicate a worse outcome.
Modified Fatigue Impact Scale | 12 Weeks
  The effect of fatigue on cognitive, physical, and psychosocial functioning will be measured with the modified fatigue impact scale. The minimum score is 0, the maximum score is 36, and higher scores indicate a worse outcome.
Connor Davidson Resilience Scale 10 | 12 Weeks
  Resilience will be measured on the Connor Davidson Resilience Scale 10. The minimum score is 0, the maximum score is 40, and higher scores indicate a better outcome.
Lower Extremity Function Scale | 12 Weeks
  Ability to perform every day tasks will be measured on the Lower Extremity Function Scale. The minimum score is 0, the maximum score is 80, and lower scores indicate worse outcomes.
Capability, Opportunity, Motivation, Behavior (COM-B) Survey | 12 Weeks
  Capability, opportunity, and motivation for behavior change will be measured on the COM-B survey. The minimum score is 0, the maximum score is 60, and higher scores indicate better outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Puneeta Tandon, Principal Investigator — University of Alberta
Locations (1):
- University of Alberta, Edmonton, Alberta, Canada